CLINICAL TRIAL: NCT03147885
Title: A Phase 1b/2 Investigator Initiated Study of RCHOP in Combination With Selinexor (KPT-330) in B Cell Non-Hodgkin's Lymphoma
Brief Title: Selinexor Plus Combination Chemotherapy in Treating Patients With Advanced B Cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dipenkumar Modi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-125; P30CA022453 (NIH)
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B-Cell Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Extranodal Marginal Zone Lymphoma; Recurrent Follicular Lymphoma; Recurrent Indolent Adult Non-Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Waldenstrom Macroglobulinemia; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Extranodal Marginal Zone Lymphoma; Refractory Follicular Lymphoma; Refractory Mantle Cell Lymphoma; Stage III Non-Hodgkin Lymphoma; Stage IV Non-Hodgkin Lymphoma; Transformed Recurrent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Lymphoma, Non-Hodgkin | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (selinexor, RCHOP) (Experimental): Patients will receive selinexor PO on days 1, 8, and 15 of a 21 week cycle. RCHOP will be given at standard dosing every 21 days. In the phase 1 part there is dose escalation for Selinexor in a 3+3 design. Treatment will be given for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with partial response or better will receive maintenance selinexor PO on days 1, 8, 15, and 22 every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Given PO
  Other Names: CRM1 Nuclear Export Inhibitor KPT-330; KPT-330; Selective Inhibitor of Nuclear

SUMMARY:
This phase Ib/II trial is aimed at studying the combination of a drug named Selinexor (selective inhibitor of nuclear export) in combination with standard therapy for B cell Non-Hodgkin's lymphoma called R-CHOP. The investigators will establish maximum tolerated dose of Selinexor in combination with RCHOP and also study the efficacy of this combination for therapy of B cell Non-Hodgkin's lymphoma. Giving Selinexor plus chemotherapy may work better in treating patients with B cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
The study will be done in two phases namely phase 1B and phase 2.

In the phase 1B component the investigators intend to enroll patients in a 3+3 dose escalation design. Newly diagnosed indolent and diffuse large cell lymphomas as well as relapsed/refractory indolent B cell lymphomas are eligible for enrollment in the phase 1 component. The primary end-point for this component would be to establish the recommended phase 2 dose (RP2D) for Selinexor in combination with standard dose RCHOP chemotherapy.

In the phase 2 part of the study the investigators will use recommended phase 2 dose of Selinexor plus standard dose RCHOP combination to treat newly diagnosed DLBCL patients with the primary end-point being 2 year Progression free survival.

Maintenance Phase: Patients with Follicular Lymphoma and Diffuse Large B cell lymphoma able to achieve PR or better at the end of therapy scan will be put on maintenance Selinexor for a total of one year. The dose of Selinexor in the maintenance phase would be similar to the last dose used for that particular patient in the treatment phase 1 or 2.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 Part: Patients with pathologically confirmed advanced stage B-cell NHL (Ann Arbor stage 3 or 4) for whom R-CHOP is considered appropriate therapy; newly diagnosed DLBCL, newly diagnosed low grade B cell NHL, and previously treated low grade B cell NHL patients in first relapse after a prior treatment with non-anthracycline containing chemotherapy are allowed; double hit and transformed diffuse large B cell lymphoma are allowed

  * Allowed low grade B cell lymphomas will include follicular lymphoma any grade, marginal zone lymphoma including mucosa-associated lymphoid tissue (MALT) lymphoma, indolent mantle cell lymphoma and Waldenstrom's macroglobulinemia
* Phase 2 Part: Patients with pathologically confirmed newly diagnosed diffuse large B cell lymphoma (Ann Arbor stage 3 or 4); newly diagnosed double hit and transformed diffuse large B cell lymphoma are allowed
* Patients must have measurable disease, defined as at least one lesion above and below the diaphragm or stage 4 disease that can be accurately measured in at least one dimension; lymph nodes should be considered abnormal if the long axis is > 1.5 cm, regardless of the short axis
* Allowed prior therapy:

  * Newly diagnosed DLBCL and low grade B cell lymphoma: No prior therapy is allowed except steroids equivalent to maximum of prednisone 20 mg once daily for maximum of seven days prior to registration
  * Relapsed/refractory low grade B cell lymphoma (only allowed in phase I): A minimum and maximum of one line of prior non-anthracycline containing therapy is allowed; prior localized radiation therapy is not considered a line
  * For patients who have had prior chemotherapy or immunotherapy, at least 2 weeks must have elapsed between last dose and initial dose of RCHOP-selinexor; for patients treated with radio-immunotherapy, at least 12 weeks
* All races and ethnic groups are eligible for this trial
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months
* Premenopausal female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential; acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal; for both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with DLBCL who have received chemotherapy or immunotherapy (except one week of steroids as described above) at any time point in the past for therapy of the DLBCL; patients with low grade B cell lymphomas who have received more than one prior line of chemotherapy or any anthracycline-containing therapy in the past for their low grade B cell lymphoma; localized radiation therapy does not count as a line of therapy
* Patients who are receiving any other investigational agents
* Patients with known brain metastases are excluded
* History of severe allergic reactions (as determined by treating physician) attributed to the drugs being used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congestive heart failure (New York Heart Association [NYHA] class >= 3 or left ventricular ejection fraction < 45%), unstable angina pectoris, myocardial infarction within the last 3 months, clinically significant cardiac arrhythmia (i.e., ventricular tachycardia on anti-arrhythmia are excluded; 1st degree atrioventricular [AV] block or asymptomatic left anterior fascicular block [LAFB]/right bundle branch block [RBBB] permissible), or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and lactating women are excluded
* Human immunodeficiency virus (HIV)-positive patients regardless of treatment are excluded; patients with evidence of active hepatitis B and hepatitis C infection with positive real time polymerase chain reaction (qPCR) are also excluded but patients with prior exposure to hepatitis B or C with negative qPCR are allowed
* Patients with severe intolerance to glucocorticoids
* Major surgery within 2 weeks of first dose of study drug
* Patients who are unable to swallow tablets, patients with malabsorption syndrome, or any other gastrointestinal (GI) disease or GI dysfunction that could interfere with absorption of study treatment
* Absolute neutrophil count (ANC) < 1500 cells/mm^3
* Platelet count < 100,000/mm^3
* Serum bilirubin > 1.5 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome: total bilirubin of > 3 x ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 times ULN
* Estimated creatinine clearance of < 30 mL/min, calculated using the formula of Cockroft and Gault

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of selinexor in combination with RCHOP chemotherapy defined as =< 1/6 patients experience a dose limiting toxicity (Phase Ib) | Up to 21 days
  Toxicity grading in both phase 1b and phase 2 parts will be done based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 guidelines. Toxicity data will be collected at least weekly during the course of treatment. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Progression-free survival (PFS) for patients with newly diagnosed DLBCL treated with RCHOP-selinexor combination (Phase II) | From baseline to disease progression or death from any cause, assessed up to 2 years
  PFS will be described with Kaplan-Meier curves and estimated medians with 95% confidence intervals.

SECONDARY OUTCOMES:
CR of patients with newly DLBCL treated with selinexor and RCHOP | Up to 2 years
  Response rates will be estimated as proportions with 95% Wilson confidence intervals.
PR of patients with newly diagnosed DLBCL treated with selinexor and RCHOP | Up to 2 years
  Response rates will be estimated as proportions with 95% Wilson confidence intervals.
SD of patients with newly diagnosed DLBCL treated with selinexor and RCHOP | Up to 2 years
  Response rates will be estimated as proportions with 95% Wilson confidence intervals.
ORR (CR and PR) of patients with newly diagnosed DLBCL treated with selinexor and RCHOP | Up to 2 years
  Response rates will be estimated as proportions with 95% Wilson confidence intervals.
OS of patients with newly diagnosed DLBCL treated with RCHOP-selinexor combination | Baseline to date of death, assessed up to 2 years
  OS will be described with Kaplan-Meier curves and estimated medians with 95% confidence intervals.
Change in CRM1/XPO-1 activity expression assessed in tissue by polymerase chain reaction (PCR) | Baseline and at 48-72 hours after cycle 1 day 1
  Difference in the CRM-1 activity by PCR in the tumor tissue and peripheral blood samples obtained at baseline and at 48-72 hours after cycle 1 day1 of therapy.
Change in CRM1/XPO-1 activity expression assessed in tissue by immunohistochemistry (IHC) | Baseline and at 48-72 hours after cycle 1 day 1
  Difference in the CRM-1 activity by IHC in the tumor tissue and peripheral blood samples obtained at baseline and at 48-72 hours after cycle 1 day1 of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dipenkumar Modi, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seymour EK, Khan HY, Li Y, Chaker M, Muqbil I, Aboukameel A, Ramchandren R, Houde C, Sterbis G, Yang J, Bhutani D, Pregja S, Reichel K, Huddlestun A, Neveux C, Corona K, Landesman Y, Shah J, Kauffman M, Shacham S, Mohammad RM, Azmi AS, Zonder JA. Selinexor in Combination with R-CHOP for Frontline Treatment of Non-Hodgkin Lymphoma: Results of a Phase I Study. Clin Cancer Res. 2021 Jun 15;27(12):3307-3316. doi: 10.1158/1078-0432.CCR-20-4929. Epub 2021 Mar 30. PMID 33785483